CLINICAL TRIAL: NCT06502379
Title: A Phase I Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, and Pharmacokinetics of AZD8965 Following Single and Multiple Ascending Dose Administration to Healthy Participants (Including Japanese and Chinese Participants) and an Open-label Cohort to Assess the Effect of Food on the Pharmacokinetics of AZD8965 in Healthy Participants
Brief Title: A Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of AZD8965 in Healthy Participants (Including Japanese and Chinese Participants) and an Open-label Cohort to Assess the Effect of Food on the Pharmacokinetics of AZD8965 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D6960C00001
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: Idiopathic Pulmonary Fibrosis; Lung disease; Pharmacokinetics; Food Effect
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part 1: SAD Cohort 1 - AZD8965 (Dose 1) (Experimental): Participants will receive a single dose of AZD8965 (Dose 1) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 1: SAD Cohort 2 - AZD8965 (Dose 2) (Experimental): Participants will receive a single dose of AZD8965 (Dose 2) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 1: SAD Cohort 3 - AZD8965 (Dose 3) (Experimental): Participants will receive a single dose of AZD8965 (Dose 3) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 1: SAD Cohort 4 - AZD8965 (Dose 4) (Experimental): Participants will receive a single dose of AZD8965 (Dose 4) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 1: SAD Cohort 5 - AZD8965 (Dose 5) (Experimental): Participants will receive a single dose of AZD8965 (Dose 5) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 2: MAD Cohort 1 - AZD8965 (Dose 1) (Experimental): Participants will receive multiple doses of AZD8965 (Dose 1) or matching placebo to AZD8965 from Day 1 to Day 8.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 2: MAD Cohort 2 - AZD8965 (Dose 2) (Experimental): Participants will receive multiple doses of AZD8965 (Dose 2) or matching placebo to AZD8965 from Day 1 to Day 8.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 2: MAD Cohort 3 - AZD8965 (Dose 3) (Experimental): Participants will receive multiple doses of AZD8965 (Dose 3) or matching placebo to AZD8965 from Day 1 to Day 8.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 3A: SAD Cohort 1 (Japanese) - AZD8965 (Dose 1) (Experimental): Japanese participants will receive a single dose of AZD8965 (Dose 1) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 3A: SAD Cohort 2 (Japanese) - AZD8965 (Dose 2) (Experimental): Japanese participants will receive a single dose of AZD8965 (Dose 2) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 3A: SAD Cohort 3 (Chinese) - AZD8965 (Dose 1) (Experimental): Chinese participants will receive a single dose of AZD8965 (Dose 1) or matching placebo to AZD8965 on Day 1.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 3B: Single and multiple ascending dose (SMAD) Cohort 1 (Japanese) - AZD8965 (Dose 1) (Experimental): Japanese participants will receive a single dose of AZD8965 (Dose 1) or matching placebo to AZD8965 on Day 1, followed by multiple doses of AZD8965 or matching placebo from Day 3 until Day 9.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 3B: SMAD Cohort 2 (Chinese) - AZD8965 (Dose 1) (Experimental): Chinese participants will receive a single dose of AZD8965 (Dose 1) or matching placebo to AZD8965 on Day 1, followed by multiple doses of AZD8965 or matching placebo from Day 3 until Day 9.
  Interventions: Drug: AZD8965; Other: Placebo
- Part 4: Food Effect Cohort - AZD8965 (Experimental): Participants will receive 2 single dose treatments of AZD8965 [following an overnight fast of at least 10 hours in a fasted state or a fed state (after a high fat meal)].
  Interventions: Drug: AZD8965

INTERVENTIONS:
Drug: AZD8965 — AZD8965 will be administered orally.
Other: Placebo — Placebo will be administered orally.
  Arms: Part 1: SAD Cohort 1 - AZD8965 (Dose 1); Part 1: SAD Cohort 2 - AZD8965 (Dose 2); Part 1: SAD Cohort 3 - AZD8965 (Dose 3); Part 1: SAD Cohort 4 - AZD8965 (Dose 4); Part 1: SAD Cohort 5 - AZD8965 (Dose 5); Part 2: MAD Cohort 1 - AZD8965 (Dose 1); Part 2: MAD Cohort 2 - AZD8965 (Dose 2); Part 2: MAD Cohort 3 - AZD8965 (Dose 3); Part 3A: SAD Cohort 1 (Japanese) - AZD8965 (Dose 1); Part 3A: SAD Cohort 2 (Japanese) - AZD8965 (Dose 2); Part 3A: SAD Cohort 3 (Chinese) - AZD8965 (Dose 1); Part 3B: SMAD Cohort 2 (Chinese) - AZD8965 (Dose 1); Part 3B: Single and multiple ascending dose (SMAD) Cohort 1 (Japanese) - AZD8965 (Dose 1)

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics (PK) of AZD8965 via single and multiple ascending doses in healthy participants (including Japanese and Chinese participants), and to assess the effect of food on the safety, tolerability, and PK of orally administered AZD8965.

DETAILED DESCRIPTION:
This is a first in human single and multiple ascending dose study. The study consists of 4 parts: Part 1 (single ascending dose [SAD]), Part 2 (multiple ascending dose [MAD]), Part 3A (Japanese and Chinese SAD), Part 3B (Japanese and Chinese combined SAD and MAD), and Part 4 (Food Effect).

Each study part includes a 28-day screening period and a residential period during which participants will be resident at the Clinical Unit from the day before study intervention administration (Day -1) until at least 48-72 hours after the study intervention administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants (including Japanese and Chinese participants) with suitable veins for cannulation or repeated venipuncture.
* All females of childbearing potential must have a negative pregnancy test at the Screening Visit (serum) and on admission (urine) to the Clinical Unit.
* All females of childbearing potential must not be lactating and if heterosexually active must agree to use an approved method of highly effective contraception with low user dependency and their non-sterilized male partners must use a condom, to avoid pregnancy from the time of first administration of study intervention until 20 days after the last dose of study intervention. Females must not use hormonal contraceptives or hormone replacement therapy during the study.
* Females of non-childbearing potential must be confirmed at the Screening Visit by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months following cessation of all exogenous hormonal treatments and without an alternative medical cause and the follicle stimulating hormone (FSH) level is in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy. Tubal ligation is not acceptable.
* Sexually active fertile male participants with partners of childbearing potential must adhere to the specified contraception methods from the time of first administration of study intervention administration until 20 days after the last dose of study intervention.
* Have a body mass index (BMI) between 18 and 30 kilogram (kg)/square meter (m2) inclusive and weigh at least 45 kg.

Part 3A and Part 3B (Japanese Participants)

* Healthy Japanese participants are eligible based on meeting all of the following:

  1. Born in Japan
  2. Have 2 Japanese biological parents and 4 Japanese grandparents.
  3. Did not live outside Japan for more than 10 years at the time of Screening. Part 3A and Part 3B (Chinese Participants)
* Healthy Chinese participants. Participants of Chinese ancestry are eligible based on meeting all of the following:

  1. Born in mainland China, Hong Kong, Macau, or Taiwan
  2. Have 2 Chinese biological parents and 4 Chinese grandparents as confirmed by the interview.
  3. Did not live outside China for more than 10 years at the time of Screening.

Exclusion Criteria:

* History of any clinically important disease or disorder which may either put the participant at risk or influence the results or the participant's ability to participate in the study.
* Chronic or ongoing gastrointestinal, respiratory, hepatic, renal disease, pancreatic disease, diabetes mellitus, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Chronic or ongoing neurological disorder, any clinically important past or ongoing psychiatric disorder which may confound assessment of the potential neurologic effects of this product.
* Participants with a history of hypertension or cardiovascular disease.
* Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of study intervention.
* Participant with chronic infections (e.g., urinary tract infection) or who are at increased risk of infection (e.g., surgery, trauma, severe dental disease, or significant infection).
* Participants with a known or suspected defect in the function of the urea cycle, or with family history of a urea cycle disorder in one or more biological relative.
* Any abnormal laboratory values and vital signs.
* Ongoing acquired or inherited immunodeficiency disorders, including but not limited to human immunodeficiency virus (HIV) or common variable immunodeficiency, or the participant is taking immune replacement therapy.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8965.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 147 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 3A: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | SAEs: From Screening (Day -28) to 5 weeks; AEs: From Day 1 to 5 weeks
  To assess the safety and tolerability of AZD8965 following oral administration of single ascending doses to healthy participants.
Parts 2 and 3B: Number of participants with AEs and SAEs | SAEs: From Screening (Day -28) to 8 weeks; AEs: From Day 1 to 8 weeks.
  To assess the safety and tolerability of AZD8965 following oral administration of multiple ascending doses to healthy participants.
Part 4: Maximum observed drug concentration (Cmax) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Area under concentration-time curve from time 0 to infinity (AUCinf) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Time to reach maximum observed concentration (tmax) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Partial area under the concentration-time curve from time t1 to time t2 [AUC(t1-t2)] | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Terminal elimination half-life (t½λz) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Mean Residence Time (MRTinf) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Apparent total body clearance (CL/F) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Apparent volume of distribution based on the terminal (Vz/F) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Accumulation ratio for AUC (Rac AUC) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Accumulation ratio for Cmax (Rac Cmax) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | From Day 1 (pre-dose) to Day 5
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | From Day 1 (pre-dose) to Day 5
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Relative bioavailability calculated as test AUC/reference AUC (Frel AUC) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Relative bioavailability calculated as test Cmax/reference Cmax (Frel Cmax) | From Day 1 (pre-dose) to Day 7 (72-hour post dose)
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.
Part 4: Renal clearance (CLR) | From Day 1 (pre-dose) to Day 5
  To assess the effect of a high fat meal compared to fasting conditions on the PK of active drug and pro-drug following oral administration of AZD8965 in healthy participants.

SECONDARY OUTCOMES:
Parts 1, 2, 3A and 3B: Maximum observed drug concentration (Cmax) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Area under concentration-time curve from time 0 to infinity (AUCinf) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Time to reach maximum observed concentration (tmax) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Partial area under the concentration-time curve from time t1 to time t2 [AUC(t1-t2)] | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Terminal elimination half-life (t½λz) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Mean Residence Time (MRTinf) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Apparent total body clearance (CL/F) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Apparent volume of distribution based on the terminal (Vz/F) | Parts 1 and 3A: From Day 1 (pre-dose) to Day 4 (72-hour post dose); Parts 2 and 3B: From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Individual and cumulative amount of unchanged drug excreted into urine from time t1 to time t2 [Ae(t1-t2)] | Parts 1 and 3A: Up to Day 2; Parts 2 and 3B: Days 1, 2, 8, 9
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Individual and cumulative percentage of dose excreted unchanged in urine from time t1 to time t2 [fe(t1-t2)] | Parts 1 and 3A: Up to Day 2; Parts 2 and 3B: Days 1, 2, 8, 9
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 1, 2, 3A and 3B: Renal clearance (CLR) | Parts 1 and 3A: Up to Day 2; Parts 2 and 3B: Days 1, 2, 8, 9
  To characterize the PK of active drug and pro-drug following oral administration of single and multiple ascending doses of AZD8965 in healthy participants.
Parts 2 and 3B: Area under concentration-time curve in the dosing interval (AUCtau) | From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of multiple ascending doses of AZD8965 in healthy participants.
Parts 2 and 3B: Accumulation ratio for AUC (Rac AUC) | From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of multiple ascending doses of AZD8965 in healthy participants.
Parts 2 and 3B: Accumulation ratio for Cmax (Rac Cmax) | From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of multiple ascending doses of AZD8965 in healthy participants.
Parts 2 and 3B: Temporal Change Parameter (TCP) | From Day 1 (pre-dose) to Day 10 (48-hour post dose)
  To characterize the PK of active drug and pro-drug following oral administration of multiple ascending doses of AZD8965 in healthy participants.
Part 4: Number of participants with AEs and SAEs | SAEs: From Screening (Day -28) to 6 weeks; AEs: From Day 1 to 6 weeks
  To assess the safety and tolerability of AZD8965 under fasted and fed (after intake of a high fat meal) conditions in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/